CLINICAL TRIAL: NCT02983396
Title: The Accuracy of the Mini RELF Device Relative to the 12 Lead ECG for the Diagnosis of an Acute Coronary Artery Occlusion in Patients With Coronary Artery Disease.
Brief Title: The Accuracy of the Mini RELF Device for the Diagnosis of an Acute Coronary Artery Occlusion.
Acronym: RELF IIa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UniversityGhent
Record Dates: First submitted 2016-10-25; First posted 2016-12-06 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Chest Pain; ST Elevation Myocardial Infarction
Keywords: RELF method; Medical device; Admission delay
MeSH Terms: conditions — Chest Pain; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- no transmural ischemia (NTI) and transmural ischemia (TI) (Experimental): Case cross-over from "no transmural ischemia (NTI)" to "transmural ischemia at 60 s coronary occlusion during elective coronary angioplasty (TI)"
  Comparison of diagnostic accuracy of standard 12-lead ECG versus Mini RELF device for detection of transmural ischemia.
  Interventions: Device: Diagnostic accuracy of Mini Relf Device

INTERVENTIONS:
Device: Diagnostic accuracy of Mini Relf Device — Evaluation of the Mini Relf Device when it is applied on daily basis at home and during coronary angioplasty at 60 second acute coronary occlusion angioplasty

SUMMARY:
Patient delay in seeking medical attendance for symptoms of acute ST elevation myocardial infarction (STEMI) is the major obstacle to reduce the current mortality from acute coronary syndromes. The Mini RELF device is a hand held self applicable device intended to detect on an individual basis an elevation of the ST segment that is indicative for an acute coronary occlusion. The investigators aim to evaluate the accuracy of Mini RELF device when it is self-applied on a daily basis by patients with coronary artery disease.

DETAILED DESCRIPTION:
The increasing availability of small hand held medical devices is a novel opportunity to develop a tool that guides patients through the decision-taking processes of seeking medical attendance during symptoms suggestive of acute myocardial infarction. The cornerstone of early diagnosis, risk stratification and treatment is the presence of ST segment elevation during symptoms suggestive of STEMI. Therefore, a hand held medical device that can detect ST segment elevation with high sensitivity and specificity could be a breakthrough in the further reduction of fatality from acute myocardial infarction. A number of conditions of the tool must be fulfilled to allow save use with a low threshold in the general population. Most important is the accuracy to detect any new ST segment elevation related to an acute artery occlusion. For more than 30 years the 12-lead ECG is the gold standard for detection of ST elevation. However, acute coronary occlusions of a posterior or lateral segment are not always detected by the gold standard. Moreover, in the very early phase of acute coronary occlusion, the accuracy 12 lead ECG is inadequate.

In a previous study "Diagnostic accuracy of a novel method for detection of acute transmural myocardial ischemia based upon a self-applicable 3-lead configuration" the investigators developed and validated a sensitive and specific 3-lead ECG method (RELF method). The method includes a new lead configuration and a new algorithm to analyze the ECG recordings based on an intra-individual comparisons of ST levels. In summary, a 3-lead recording from a healthy subject or from a patient with an acute coronary occlusion is compared automatically to one or more previous reference recordings from the same individual. The individualized ST shift is used as a decision variable to detect or reject an acute coronary artery occlusion. The RELF method was more accurate then the simultaneously applied 12-lead ECG which had a lower sensitivity and specificity. In that study all recordings were performed by a sophisticated ECG recording system. The RELF method is designed to be applicable also by small hand held ECG devices such as the self-applicable Mini RELF device.

In the current study the investigators aim to evaluate the accuracy of Mini RELF device relative to the 12 lead ECG when the device is self-applied on a daily basis by patients with coronary artery disease. In a parallel study (RELF IIb) the investigators aim to evaluate the specificity of the RELF method when it is self-applied by healthy subjects who are representative for future users of the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an appointment for an elective coronary angioplasty.

Exclusion Criteria:

* Patients with coronary artery bypass grafts.
* Patients with implanted pacemaker or ICD.
* Patients who remain hospitalized until the planned angioplasty.
* Patient who are unfamiliar with use of smart phone. The test question "did you use by yourself a smart phone to make a telephone call in the last 4 weeks" should be answered by yes.
* Patients who cannot tolerate repetitive applications of standard skin electrodes on the chest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
The accuracy (Area under the sensitivity-aspecificity curve) of Modus RELF-2 (The orthonormalized ST shift vector magnitude) | One week after coronary angioplasty
  The sensitivity and specificity of the orthonormalized ST shift vector magnitude during occlusion compared to the sensitivity and specificity of the 12 lead ECG.

SECONDARY OUTCOMES:
The accuracy (Area under the sensitivity-aspecificity curve) of Modus RELF-3 | One week after coronary angioplasty
  The sensitivity and specificity of the intraindividual orthonormalized ST shift vector magnitude
The accuracy (Area under the sensitivity-aspecificity curve) of Modus RELF-1 (The gender specific orthonormalized ST vector magnitude) and of Modus RELF-3 (The intra-individual orthonormalized ST shift vector magnitude). | One week after coronary angioplasty
  The sensitivity and specificity of the gender specific orthonormalized ST vector magnitude and the intra-individual orthonormalized ST shift vector magnitude during occlusion compared to the sensitivity and specificity of the 12 lead ECG.
Number of participants with symptoms of contact dermatitis in the thoracic device-skin contact area. | One week after coronary angioplasty
  Contact dermatitis is defined by the clinical presence of redness or itching or blistering delineated in the thoracic device-skin contact area during at least one of the three clinical visits in the study participation period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gheeraert, Professor, Study Chair — University Ghent, Belgium
Locations (3):
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Jan Brugge, Bruges
  - University Hospital Ghent, Ghent
  - AZ Sint Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Heuverswyn F, De Buyzere M, Coeman M, De Pooter J, Drieghe B, Duytschaever M, Gevaert S, Kayaert P, Vandekerckhove Y, Voet J, El Haddad M, Gheeraert P. Feasibility and performance of a device for automatic self-detection of symptomatic acute coronary artery occlusion in outpatients with coronary artery disease: a multicentre observational study. Lancet Digit Health. 2019 Jun;1(2):e90-e99. doi: 10.1016/S2589-7500(19)30026-3. Epub 2019 May 23. PMID 33323233